CLINICAL TRIAL: NCT05628636
Title: A Phase 1, Open-label Study to Evaluate the Tolerability of 21 Days of Treatment With the AC-OLE-01-VA Formulation of Tricaprilin Under Different Dosing Conditions in Healthy Participants
Brief Title: AC-OLE-01-VA Tolerability Study in Healthy Participants Under Different Dosing Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AC-22-031
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Days 1-3: 5 g BID 4-6: 10 g BID 7-9: 15 g BID 10-21: 20 g BID
  Interventions: Drug: AC-OLE-01-VA
- Arm 2 (Experimental): Days 1-3: 10 g BID 4-6: 10 g BID 7-9: 10 g BID 10-21: 20 g BID
  Interventions: Drug: AC-OLE-01-VA
- Arm 3 (Experimental): Days 1-3: 15 g TID 4-6: 10 g TID 7-9: 10 g TID 10-21: 15 g TID
  Interventions: Drug: AC-OLE-01-VA

INTERVENTIONS:
Drug: AC-OLE-01-VA — formulation of tricaprilin

SUMMARY:
This is an open-label, 3-arm study to compare tolerability of three different titration and dosing schedules of the AC-OLE-01-VA formulation of tricaprilin.

Following a screening of up to 28 days, eligible participants will be initially randomised to one of 2 arms (Arm 1 or Arm 2). Arms 1 and 2 will be completed in advance of Arm 3 with all subsequent participants allocated to Arm 3.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy (in the opinion of the Investigator) as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight ≥45 kg and body mass index (BMI) within the range 18.0 - 32.0 kg/m2 (inclusive).

Exclusion Criteria:

* History of, or current gastrointestinal (GI) conditions constituting a risk when taking the study treatment; or interfering with the interpretation of data, based on the Investigator's judgement.
* Participants on a ketogenic diet, low-fat diet or actively using medium chain triglycerides, ketone esters, or other ketogenic products within 3 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Ratings of discomfort of the adverse events nausea, dyspepsia, abdominal pain, abdominal distension, diarrhoea | 21 days
  Discomfort rating from 0 (no discomfort) to 4 (severe discomfort)
Incidence of adverse events | 21 days
  Adverse event incidence will be tabulated Adverse event incidence will be tabulated Adverse event incidence will be tabulated

CONTACTS AND LOCATIONS:
Locations (1):
- RDC Clinical, Newstead, Queensland, Australia